CLINICAL TRIAL: NCT05621187
Title: BIO|MASTER.Pamira Study
Brief Title: Post Market Clinical Follow-up Study for the Pamira ICD Lead Family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TA117
Record Dates: First submitted 2022-11-07; First posted 2022-11-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Tachyarrhythmia
MeSH Terms: conditions — Heart Failure; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other)
  Interventions: Device: Pamira ICD lead family

INTERVENTIONS:
Device: Pamira ICD lead family — Implantation, measurements and follow-up schedule

SUMMARY:
Confirm clinical safety and performance of the Pamira lead to support the regulatory post market strategy in Europe and other regions and validating promotional claims by

* demonstrating clinical safety
* evaluating performance based on sensing and pacing assessment
* collecting additional data of interest to assess other aspects such as the handling and usability

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD or CRT-D therapy according to clinical guidelines
* Planned for de novo implantation of a BIOTRONIK ICD or CRT-D in combination with Pamira
* Ability to understand the nature of the study and willingness to provide written informed consent
* Ability and willingness to perform all follow-up visits at the study site
* Ability and willingness to use the CardioMessenger and acceptance the BIOTRONIK Home Monitoring® concept

Exclusion Criteria:

* Mechanical tricuspid valve prosthesis or a severe tricuspid valve disease
* Known Dexamethasone acetate intolerance
* Cardiac surgical post-implantation procedure planned within 12 months (including interventional procedures like ablation, valve replacement, heart transplant etc.)
* Less than 18 years old
* Pregnant or breast feeding
* Participating in another interventional clinical investigation
* Life-expectancy less than 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Pamira lead related SADE-d free rate at 6 months after implantation | 6 months

SECONDARY OUTCOMES:
1a and b: Pamira lead related SADE-d free rate at 3 and 12 months after implantation | 3 months, 12 months
2a and 2b: Rate of appropriate right ventricular sensing at the 6- and 12-month follow-up | 6 months, 12 months
3a and 3b: Rate of appropriate right ventricular pacing at the 6- and 12-month follow-up | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Deneke, Prof., Principal Investigator — RHÖN-KLINIKUM Campus Bad Neustadt, Germany
Locations (23):
- John Hunter Hospital, New Lambton Heights, New South Wales, Australia
- Medizinische Universität Graz, Graz, Styria, Austria
- Belgium (2):
  - UZ Brussels, Jette
  - UZ Leuven Gasthuisberg, Leuven
- Germany (11):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau bei Berlin, Brandenburg
  - St. Marienkrankhaus Klinikum Westmünsterland GmbH, Ahaus, North Rhine-Westphalia
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden, Saxony
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg, Saxony-Anhalt
  - Klinikum Dorothea Christiane Erxleben Quedlinburg, Quedlinburg, Saxony-Anhalt
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - SRH Zentralklinikum Suhl GmbH, Suhl, Thuringia
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
- Hungary (3):
  - State Hospital of Cardiology, Balatonfüred
  - Semmelweis University, Budapest
  - The University of Pécs, Pécs
- Israel (3):
  - Assuta Medical Center, Ashdod
  - Soroka Medical Center, Beersheba
  - Shaare Zedek MC, Jerusalem
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Stredoslovenský ústav srdcových a cievnych chorôb, a.s. (SÚSCCH, a.s.), Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: No